CLINICAL TRIAL: NCT00458055
Title: Treatment Study for Severe High-Density Lipoprotein Deficiency
Brief Title: High-Density Lipoprotein (HDL) Treatment Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Jacques Genest MD, McGill University Hospital Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUHC-RI 0906
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Coronary Arteriosclerosis; Hypoalphalipoproteinemias; Genetic Diseases, Inborn
Keywords: Lipid lowering agents; Drug treatment; Statin; Fibrate; Niacin; Cellular cholesterol efflux
MeSH Terms: conditions — Coronary Artery Disease; Hypoalphalipoproteinemias; Genetic Diseases, Inborn | interventions — Atorvastatin; Fenofibrate; Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Atorvastatin; Fenofibrate; Niacin — Atorvastatin 20 mg; Fenofibrate 200 mg; Niacin 2g used sequentially for 8 weeks, after 4 weeks washout.
  Other Names: Lipotor; Tricor; Niaspan

SUMMARY:
A low level of plasma high-density lipoprotein (HDL) cholesterol, "the good cholesterol", is the most common lipid abnormality observed in patients with a premature atherosclerotic cardiovascular disease. HDL carry excess cholesterol from peripheral tissues to the liver to be metabolized or excreted, a process known as reverse cholesterol transport.

Epidemiological studies have shown an inverse correlation between plasma levels of HDL cholesterol and the risk of cardiovascular disease. An increase in plasma HDL cholesterol levels by 1 mg/dL may reduce the risk of cardiovascular disease by 2 to 3%. The standard care of treatment for a low level of HDL cholesterol is: 1) lifestyle modifications including exercise, smoking cessation, weight control, moderate alcohol intake and decreased dietary fat intake - all patients are encouraged to follow these lifestyle modifications; 2) medications which can raise HDL cholesterol.

Currently used medications to treat lipid disorders can increase, in some extent, HDL cholesterol. These include niacin (vitamin B3), fibric acid derivatives (fibrates) and statins. However there is no data on the effect of these medications on severe cases of HDL deficiency. This project aims to determine whether currently available medications, used in standard medical practice for the treatment of lipoprotein disorders, can substantially increase HDL cholesterol in severe cases of HDL deficiencies.

DETAILED DESCRIPTION:
Objective and rationale. We have collected, in the past 15 years, a large group of patients with familial HDL cholesterol deficiency. In approximately 25% of index probands in our family studies, the genetic basis of HDL deficiency is identified at the molecular level. Approximately 20% of our severe HDL cholesterol deficient patients have mutations within the ABCA1 gene, while mutations at the apoA-I and SMPD1 genes have also been identified. In the present study, we wish to determine whether conventional lipid-regulating medication can substantially increase HDL cholesterol in patients with severe HDL deficiency. Anecdotal reports from our clinic suggest that patients with ABCA1 mutations do not respond to currently available medication; this will be more thoroughly ascertain in this protocol. In addition, examining patients with other genetic HDL deficiencies and familial forms (gene not yet identified) will provide insight on the treatment options for these patients. We feel it is important first whether currently recommended medication can effectively raise HDL cholesterol in these patients.

Study subjects. The subjects will include patients with familial HDL deficiency (HDL cholesterol < 5th percentile for age and gender, with at least one degree relative affected) and HDL deficiency with well-defined genetic mutation. We expect approximately 20-25 patients to enter the study.

Patients will be excluded if at least one of the following criteria is present:

* Triglycerides ≥ 5 mmol/L
* Diabetes
* Severe obesity (BMI ≥ 30)
* Alcohol intake > 21 drinks/week
* Untreated disease (thyroid, hepatic or renal)

Study procedure. Patients will be treated according to current lipid treatment guidelines (McPherson R, Frohlich J, Fodor G, Genest J. Canadian Cardiovascular Society position statement: recommendations for the diagnosis and treatment of dyslipidemias and prevention of cardiovascular disease. Can J Cardiol 2006; 22:913-927) and the use of the three following medications (separately or in combination):

* Lipitor 20 mg
* Lipidil 200 mg
* Niaspan 2 g

It should be noted that all three medications are currently used to treat patients with dyslipidemia and represent the current "standard of care".

Statistics. The null hypothesis expects that no treatment effect increases HDL cholesterol by 10% in the study sample (α = 0.05 and β = 0.8). Using this study design, each patient will serve as his/her own control. Differences between baseline (B) and treatment (T) periods for each medication will be examined by sudent's t-test.

Protocol. Each treatment period will last 8 weeks; wash-out periods will last 4 weeks. Baseline values (B1-3) will be taken at the beginning of each treatment period. On-treatment values (T1-3) will be drawn at the end of each medication period. At each time B (baseline) and T (after a treatment) patient will be examined for:

* Body mass index (weight and height)
* Blood pressure
* Symptoms of ischemic heart disease
* Hepatic functions
* Myopathic symptoms

The following blood test will be performed:

* Total cholesterol
* Triglycerides
* HDL cholesterol
* LDL cholesterol
* ApoA-I, apoB
* ALT, CK

At time B1 blood will also be collected for the determination of:

* TSH
* Creatinine
* ALT
* Blood glucose

In addition, blood will be used to examine the ability of the patient's HDL and plasma to promote cellular cholesterol efflux, using an in vitro model which is well established in our laboratory. Cellular cholesterol efflux tests the efficiency of apoA-I lipidation from cells for the formation of HDL particles. This will provide a general index of the functional status of HDL particles in the body.

ELIGIBILITY:
Inclusion Criteria:

- HDL deficiency (HDL-cholesterol < 5th percentile, age and gender-matched)

Exclusion Criteria:

* Triglycerides ≥ 5 mmol/L
* Diabetes
* Severe obesity (BMI ≥ 30)
* Alcohol intake > 21 drinks/week
* Untreated disease (thyroid, hepatic or renal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
HDL cholesterol | 9 months

SECONDARY OUTCOMES:
apo AI | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Genest, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- MUHC-Royal Victoria Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] McPherson R, Frohlich J, Fodor G, Genest J, Canadian Cardiovascular Society. Canadian Cardiovascular Society position statement--recommendations for the diagnosis and treatment of dyslipidemia and prevention of cardiovascular disease. Can J Cardiol. 2006 Sep;22(11):913-27. doi: 10.1016/s0828-282x(06)70310-5. PMID 16971976
- [Background] Brewer HB Jr. High-density lipoproteins: a new potential therapeutic target for the prevention of cardiovascular disease. Arterioscler Thromb Vasc Biol. 2004 Mar;24(3):387-91. doi: 10.1161/01.ATV.0000121505.88326.d2. No abstract available. PMID 15003970
- [Background] Rubins HB, Robins SJ, Collins D, Fye CL, Anderson JW, Elam MB, Faas FH, Linares E, Schaefer EJ, Schectman G, Wilt TJ, Wittes J. Gemfibrozil for the secondary prevention of coronary heart disease in men with low levels of high-density lipoprotein cholesterol. Veterans Affairs High-Density Lipoprotein Cholesterol Intervention Trial Study Group. N Engl J Med. 1999 Aug 5;341(6):410-8. doi: 10.1056/NEJM199908053410604. PMID 10438259
- [Background] Schaefer JR, Schweer H, Ikewaki K, Stracke H, Seyberth HJ, Kaffarnik H, Maisch B, Steinmetz A. Metabolic basis of high density lipoproteins and apolipoprotein A-I increase by HMG-CoA reductase inhibition in healthy subjects and a patient with coronary artery disease. Atherosclerosis. 1999 May;144(1):177-84. doi: 10.1016/s0021-9150(99)00053-2. PMID 10381291
- [Background] Ashen MD, Blumenthal RS. Clinical practice. Low HDL cholesterol levels. N Engl J Med. 2005 Sep 22;353(12):1252-60. doi: 10.1056/NEJMcp044370. No abstract available. PMID 16177251
- [Background] Schaefer EJ, Asztalos BF. The effects of statins on high-density lipoproteins. Curr Atheroscler Rep. 2006 Jan;8(1):41-9. doi: 10.1007/s11883-006-0063-3. PMID 16455013
- See also: Cholesterol and your heart — http://www.makingtheconnection.ca/en/home
- See also: Treatment of high cholesterol — http://www.heartpoint.com/Choltreatment.html